CLINICAL TRIAL: NCT03163693
Title: The Effects of Dexmedetomidine on Cardiac Troponin I and Glycogen Phosphorylase Isoenzyme BB in Patients Undergoing Off-pump Coronary Artery Bypass Grafting
Brief Title: The Effects of Dexmedetomidine on cTnI and GP-BB in Patients Undergoing OPCABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015-NW-028
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Bypass, Off-Pump
Keywords: Dexmedetomidine; Cardiac Troponin I; Glycogen Phosphorylase Isoenzyme BB
MeSH Terms: conditions — Cardiomyopathy, Dilated, 1FF | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group dexmedetomidine (Experimental): 20 eligible patients are received 0.5ug/kg dexmedetomidine intravenously 15 minutes before surgery
  Interventions: Drug: dexmedetomidine
- Group control (Placebo Comparator): 20 eligible patients are received equal volumes normal saline intravenously 15 minutes before surgery
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: dexmedetomidine — receive dexmedetomidine 0.5 μg/kg
  Other Names: Dex
  Arms: Group dexmedetomidine
Other: normal saline — receive equal volume of normal saline
  Arms: Group control

SUMMARY:
The purpose of this study is to observe the impact of dexmedetomidine on Cardiac Troponin I and Glycogen Phosphorylase Isoenzyme BB in patients undergoing off-pump coronary artery bypass Grafting.

DETAILED DESCRIPTION:
Dexmedetomidine is a highly selective α2-adrenoceptor agonist used as a sedative or adjuvant anesthetic drug in clinical settings.From clinical observation, dexmedetomidine has been revealed to reduce the incidence of cardiovascular adverse events in patients with heart diseases during non-cardiac surgeries.Therefore, the aim of this sudy is to observe the impact of dexmedetomidine on Cardiac Troponin I and Glycogen Phosphorylase Isoenzyme BB in patients during cardiac surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing off - pump coronary artery bypass grafting
* ASA physical status III-IV
* Aged 40-70 years
* NYHA physical status II-III

Exclusion Criteria:

* Bradycardia
* Atrioventricular block
* Echocardiography suggested:LVEF <40%, LVED>65mm
* Allergic to the drugs

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change of cardiac troponin I at preoperative, postoperative，and 24 hours after surgery. | At preoperative, postoperative，and 24 hours after surgery.
  Blood samples were sampled at preoperative, postoperative，and 24 hours after surgery for the cTnI，which were analyzed by using enzyme linked immunosorbent assay (ELISA).
Change of Glycogen Phosphorylase Isoenzyme BB at preoperative, postoperative，and 24 hours after surgery. | At preoperative, postoperative，and 24 hours after surgery.
  Blood samples were sampled at preoperative, postoperative，and 24 hours after surgery for the GP-BB，which were analyzed by using enzyme linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Di, Principal Investigator — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No
safety